CLINICAL TRIAL: NCT06320756
Title: A Feasibility Study of a Digital Mental Health Intervention (Wysa in Hindi) in Improving Mental Health Distress in Adolescents and Young Adults with Type 1 Diabetes in Low Resource Settings
Brief Title: Examining the Feasibility of Wysa in Hindi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wysa (Industry)
Collaborators: Udaan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 24-WYSA-101
Record Dates: First submitted 2024-02-23; First posted 2024-03-20 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-03

CONDITIONS: Mental Health Issue; Diabetes Distress
Keywords: digital mental health
MeSH Terms: interventions — Coping Skills; Health

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial with an intervention arm and a control arm.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm: Wysa in Hindi + usual care (Experimental): The intervention arm will receive Wysa in Hindi and the usual care. Wysa in Hindi is a digital mental health intervention that combines Artificial Intelligence-led conversational chatbot support and human therapy in the Hindi language. The Artificial Intelligence (AI) chatbot acts as a companion, and understands, empathizes, and guides users through exercises grounded in cognitive behavioral therapy (CBT) techniques, written by qualified psychologists and clinicians.
  Usual care includes access to individual and bi-weekly group sessions focused on building coping, wellbeing, and motivation by the diabetes educator team.
  Interventions: Behavioral: Wysa in Hindi; Behavioral: Individual and group sessions on topics like motivation, coping, wellbeing
- Usual care arm (Active Comparator): Participants in the control group will only have access to usual care (which will remain the same as that for the intervention arm). This includes access to individual sessions and bi-weekly group sessions with the diabetes education team on motivation, wellbeing, and coping.
  Interventions: Behavioral: Individual and group sessions on topics like motivation, coping, wellbeing

INTERVENTIONS:
Behavioral: Wysa in Hindi — Wysa in Hindi is a blended digital mental health intervention
  Arms: Intervention arm: Wysa in Hindi + usual care
Behavioral: Individual and group sessions on topics like motivation, coping, wellbeing — Individual and group sessions on wellbeing, coping, and motivation with the diabetes educator team

SUMMARY:
The principal objective of this study is to investigate the feasibility of including a digital mental health intervention (Wysa in Hindi) within pre-existing usual care to support adolescents and young adults with Type 1 Diabetes (T1D) who have mild and above mental health distress (operationalized as Patient Health Questionnaire-9: 5-14 scores; or Diabetes Distress Scale-17: >2.0 mean score) with their mental health distress. This will be conducted through an exploratory randomized control study comparing Wysa in Hindi plus usual care with a control arm that just has usual care. The study further explores the effectiveness of the digital mental health intervention using the Patient Health Questionnaire (PHQ-9) and Diabetes Distress Scale (DDS-17).

DETAILED DESCRIPTION:
Participants (13-25 years) with Type1 Diabetes are invited into the study. The intervention being studied is the Wysa in Hindi app. Participants will be recruited from Udaan (a Non-Governmental Organization (NGO) supporting individuals with Type1 diabetes). They will complete baseline research procedures and be randomly allocated to one of two groups.

Participants in the intervention arm will get access to the Wysa in Hindi app as well as access to usual care (individual and group sessions on motivation, mental health, and coping). The control arm will only have access to the usual care i.e. the individual and group sessions. At the end of 2 months, participants will be invited for follow-up to complete the endline assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13-25 years
* Diagnosis of Type1 diabetes
* Access to a smartphone with internet connection
* Can read and understand Hindi
* Mental health distress as demonstrated by elevated scores on any of the scales: Mild -moderate symptoms (between 5-14 score) on Patient Health Questionnaire (PHQ-9), moderate and above diabetes distress (mean score 2.0 and higher) on the Diabetes Distress Scale (DDS-17)

Exclusion Criteria:

* Do not own or have access to a mobile device
* Are identified to have risk of harm/ suicidality (as identified on PHQ-9)
* Are currently undergoing or have received psychiatric support
* Experience any mental or physical impairments that create accessibility barriers to the use of a smartphone or access to a digital mental health intervention

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment rate (Proportion of participants who completed consent procedures) | Measured at the end of the recruitment period (3 weeks, or if recruitment is extended at the end of 2 months)
  Proportion of participants who completed consent procedures versus those who were invited to participate in the study via awareness activities.
Feasibility - Retention rate (Proportion of participants who remained enrolled within the study for the entire study duration) | Measured after the 2 month intervention during follow-up endline assessments
  Proportion of recruited participants who completed endline assessments i.e. those who remained enrolled for the study duration.
Feasibility - Wysa Engagement (Proportion of recruited participants who engaged in at least 1 interaction with the Wysa app) | Measured at the end of the 2 month intervention
  Proportion of recruited participants who interacted with Wysa at least once after onboarding to the app. Information will also collected on average numbers of days the app was used.
Feasibility - App therapist engagement rate (Proportion of recruited participants who completed at least one therapist session within the Wysa app) | Measured at the end of the 2 month intervention
  Proportion of recruited participants who completed at least one session with the therapist available on Wysa app.
Satisfaction with the app which is collected through 3 quantitative questions and 1 free text qualitative question on the app | This is collected twice; on day 2 and day 45 from onboarding on the app
  Feedback is collected through 4 questions wherein 3 questions ask participants to provide a quantitative rating of the app features' usability and satisfaction. Participants can provide ratings on a 5 point likert scale with higher ratings denoting higher satisfaction. 1 qualitative question invites participant to use free text format to provide any additional feedback. All feedback is collected twice on the app i..e. Day 2 and Day 45 from onboarding.
Therapist Satisfaction feedback collected through 3 quantitative questions and 1 free text qualitative question on the app | Collected post every therapist session during the intervention period of 2 months
  Participants provide feedback about their app therapist sessions through 3 questions asking for a quantitative rating of their satisfaction, and 1 question where participant can provide a free text response with their overall feedback. The quantitative rating is on a 5 point Likert scale with higher ratings indicating higher satisfaction. Feedback will be collected at the end of each therapist session.

SECONDARY OUTCOMES:
Change in mental health distress as measured by the Patient Health Questionnaire (PHQ-9) | Baseline assessment, and then at the 2 month follow-up endline assessment
  PHQ-9, a 9 item self report scale will be to ask about the presence of depressive symptoms. Participants are asked to rate the frequency of symptoms on a scale of 0-3. It gives a score between 0-27, with higher scores indicating more severe symptoms.
Change in mental health distress as measured by the Diabetes Distress Scale (DDS-17) | Baseline assessment, and then at the 2 month follow up assessment
  Diabetes Distress Scale (DDS-17) is a 17 item self report questionnaire on diabetes distress. Participants have to respond to how much a problem has affected their lives on a scale of 1-6. The scoring yields a mean score range between 1-6, wherein higher scores indicate higher levels of distress.

CONTACTS AND LOCATIONS:
Overall Officials: Tejaswi Shetty, M.A., Principal Investigator — Touchkin eServices Pvt. Ltd.; Archana Sarda, M.D, Principal Investigator — Udaan; Chaitali Sinha, M.A., Principal Investigator — Touchkin eServices Pvt. Ltd.
Locations (1):
- Udaan, Aurangabad, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with any external party as it does not comply with the terms of consent.

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199